CLINICAL TRIAL: NCT00003603
Title: A Randomised Study Comparing CIDEX (CCNU, Oral Idarubicin and Dexamethasone) With Melphalan and Prednisolone in Relapsed Multiple Myeloma
Brief Title: Chemotherapy Plus Steroid Therapy in Treating Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Riverside Haematology Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066676; RHG-MM97; EU-98030
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-02

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Cyclophosphamide; Dexamethasone; Idarubicin; Lomustine; Melphalan; Prednisolone

INTERVENTIONS:
Drug: cyclophosphamide
Drug: dexamethasone
Drug: idarubicin
Drug: lomustine
Drug: melphalan
Drug: prednisolone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Steroids, such as dexamethasone or prednisolone, may help relieve some of the side effects of chemotherapy. It is not yet known which regimen of chemotherapy plus steroid therapy is more effective in treating patients with multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of chemotherapy plus steroid therapy in treating patients with multiple myeloma that has recurred for the first time.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate, response duration, and survival of patients with relapsed multiple myeloma after treatment with lomustine, idarubicin, and dexamethasone vs melphalan and prednisolone.

OUTLINE: This is a randomized study. Patients are stratified according to prior autologous transplant (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral lomustine on day 1, oral idarubicin once daily on days 1-3, and oral dexamethasone twice a day on days 1-4. Treatment is repeated every 28 days for 6-9 courses in the absence of unacceptable toxicity or disease progression.
* Arm II: Patients receive oral melphalan once daily on days 1-4 and oral prednisolone twice a day on days 1-4. Treatment is repeated every 28 days for 6-9 courses in the absence of unacceptable toxicity or disease progression.

Some patients may receive oral cyclophosphamide every 7 days and oral prednisolone on alternate days for 6 weeks concurrently with chemotherapy in either treatment arm.

Quality of life is assessed at baseline, at 3, 6, 9, and 12 months, and then every 6 months thereafter.

Patients are followed until death.

PROJECTED ACCRUAL: A total of 660 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma based on at least two of the following:

  * Paraprotein in serum and/or urine
  * Greater than 10% plasma cells in bone marrow
  * Lytic bone lesions
* Measurable serum and/or urine paraprotein
* Progression from first or second stable plateau phase
* No non-secretory myeloma or plasma cell leukemia (greater than 2,000/mm^3 circulating plasma cells)
* No primary refractory disease or second or later relapse

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT/AST no greater than 2.5 times ULN

Renal:

* Creatinine less than 3.4 mg/dL

Cardiovascular:

* No clinically significant cardiac insufficiency
* No uncontrolled hypertension

Other:

* No uncontrolled diabetes mellitus
* No recent history of peptic ulceration
* HIV-1 and HIV-2 negative
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior allogeneic peripheral blood stem cell or bone marrow transplantation
* No planned future autologous transplantation unless sufficient stored stem cells available
* Prior interferon allowed if administered as maintenance of stable plateau phase
* No concurrent epoetin alfa

Chemotherapy:

* At least 3 months since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Concurrent radiotherapy for pain or to treat localized tumors allowed

Surgery:

* Not specified

Other:

* No prior participation in any clinical trial with an unlicensed product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: Diana Samson, MD, Study Chair — Hammersmith Hospitals NHS Trust
Locations (1):
- Hammersmith Hospital, London, England, United Kingdom